CLINICAL TRIAL: NCT07014124
Title: mHealth-based Motivational Counselling Integrate With a Sample of Nicotine Replacement Therapy for Fathers of Sick Children Who Smoke Cigarettes: A Pilot Randomized Controlled Trial
Brief Title: Smoking Cessation for Fathers of Sick Children
Acronym: Quit-for-Love
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Sick Children
Record Dates: First submitted 2025-01-16; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Cigarette Smoking; mHealth Intervention
Keywords: tobacco exposure; sick children; quit smoking; Nicotine replacement therapy; mHealth support; smoking fathers
MeSH Terms: conditions — Cigarette Smoking | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A 1-week free sample of NRT patch or gum will be provided to encourage quit attempt without the pressure of quitting successfully. mHealth messages will be provided to motivate and support quitting and improve the protection measured of SHS exposure for children throughout the intervention period of 3 months.
  Interventions: Behavioral: Nicotine Replacement Therapy (NRT) Sampling; Behavioral: mHealth-based motivational counselling; Behavioral: Brief cessation advice and self-help material
- Control group (Active Comparator): Participants in the control group will only receive brief advice on SHS protective measures. Self-help materials will also be provided without follow-up interventions.
  Interventions: Behavioral: Brief cessation advice and self-help material

INTERVENTIONS:
Behavioral: Nicotine Replacement Therapy (NRT) Sampling — Participants will be advised to choose the NRT according to their preferences and daily cigarette consumption. Cigarette consumption of ≤20 daily will receive the 14mg patch or 2mg gum and participants consume >20 cigarettes daily will receive the 21mg patch. An NRT use card (Appendix 6 draft) containing the instructions and potential side effects were given with a brief oral explanation. Full course of pharmacological treatment for 12-week are available in smoking cessation services. Participants requesting for additional or full course of NRT will be actively refer to the respective services as part of the Referral step in the AWARD model (Ask, Warn, Advise, Refer, and Do-it-again).
  Arms: Intervention group
Behavioral: mHealth-based motivational counselling — The mHealth intervention will be delivered via the most popular instant messaging app in Hong Kong (WhatsApp). A total of 24 messages with contents including the harms of smoking and smoke exposure for children, encouragement, benefits of quitting for children, methods of quitting, dealing with craving, and measures to reduce cigarette smoke exposure at home will be provided. The messages will be scheduled in a tapering schedule that participants will receive 5 messages in the first week, then cut down to 3 messages/week for the next 4 weeks and 1 message/week for the last 7 weeks. Using a more personalized approach, the messages will be tailored to the participants' motivation, intention to quit and other quitting patterns collected at baseline. Real-time conversations could be initiated by participants themselves, triggered by regular messages, or through prompt inquires (e.g., asking about the quitting progress).
  Arms: Intervention group
Behavioral: Brief cessation advice and self-help material — At baseline, participants will receive brief face-to-face advice on quitting smoking for the health of the children using the validated AWARD model (Ask, Warn, Advise, Refer, Do-it-again) with a print-based self-help material providing detailed information on health hazards of SHS exposure on children, methods to deal with craving and withdrawal symptoms, and measures on preventing SHS exposure for children at home.

SUMMARY:
The project aims to develop and examine the feasibility, acceptability, and preliminary effectiveness of a proactive intervention model combined brief advice, nicotine replacement therapy sampling and mHealth-based individual counselling in increasing smoking abstinence for fathers of sick children.

DETAILED DESCRIPTION:
Targeted participants are fathers of sick children who smoke daily in the past 7 days and live together with their children. The primary caregiver will be selected if both parents smoke. Participants will be recruited from pediatric wards/outpatient departments of Queen Mary Hospital (QMH), a major acute hospital in Hong Kong. The recruitment will be extended to other public hospitals if needed.

This study will be a two-arm, parallel pilot randomized trial with follow-ups at 1-, 3-, and 6-month since enrolment using standard methodology (CONSORT) to evaluate the effectiveness of the intervention. Surveys will be collected via telephone and children's saliva will be collected face-to-face at 3-months and 6-months after randomisation using Alere iScreen OFD saliva cotinine test device. Semi-structured individual telephone or face-to-face in-depth interviews will be conducted with the participants in the intervention group at 6 months follow-up to explore the participants' perception towards the intervention.

This study's clinical outcome will be biochemically validated abstinence at 3 months after randomisation. Secondary outcomes include validated abstinence at 6 months after randomisation, self-reported 7-day point prevalence abstinence (PPA), 24-hour quit attempts, and smoking reduction by at least 50% at 3 and 6 months. Incentives of HK$200 will be given to participants who report 7-day PPA at 1 month post randomisation. Additionally, incentives of HK$ 500 will be provided for the completion of each biochemical validation (a total $1000 for validation at 3- and 6-month). Such an amount can increase the response rate in our experience. Another incentive of $200 will be given to subjects completing qualitative interviews.

ELIGIBILITY:
Inclusion criteria for parents：

* Parents (mainly fathers) aged ≥18 years and smoke at least one cigarette (including alternative tobacco products) daily in the past seven days
* Living with a child aged <18 years who attended the clinic or were admitted to the pediatric ward
* Hong Kong residents able to read and communicate in Cantonese or Putonghua
* Owned a smartphone and can use an instant messaging app (e.g., WhatsApp, Facebook) Inclusion criteria for children
* Children aged <18 years who attended the clinic or were admitted to the pediatric ward
* Lives with at least one or more parents who smoke at least one cigarette (including alternative tobacco products) daily in the past seven days
* Able to provide biochemical samples (e.g. saliva) for purpose of research

Exclusion criteria for parents

* Smokers having a history of psychiatric/psychological disease or currently on regular psychotropic medications
* Smokers using smoking cessation medications or other smoking cessation services or projects Exclusion criteria for children
* Children who already have serious health diseases (e.g.chronic disease, genetic disease)
* Children who are participating in other clinical trials that may affect the results of this study
* Children who live in certain environments, such as those living in highly contaminated areas or areas with other potential disease-causing factors

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated abstinence | 3-months follow-ups
  Face-to-face biochemical validation using Alere iScreen OFD saliva cotinine test device

SECONDARY OUTCOMES:
Biochemically validated abstinence | 6-month follow-up
  Face-to-face biochemical validation using Alere iScreen OFD saliva cotinine test device
Past 7-day point prevalence abstinence (PPA) | 3-month follow-up
  Past 7-day PPA will be measured by a self-reported question: Have you ever smoked in the past 7 days?
Past 7-day point prevalence abstinence (PPA) | 6-month follow-up
  Past 7-day PPA will be measured by a self-reported question: Have you ever smoked in the past 7 days?
Smoking reduction | 3-month follow-up
  50% or above reduction in cigarette consumption compared with baseline
Smoking reduction | 6-month follow-up
  50% or above reduction in cigarette consumption compared with baseline
Use of smoking cessation services | 3-month follow-up
  Use of smoking cessation services will be measured by a self-reported question: Have you ever used smoking cessation services in the past 7 days?
Use of smoking cessation services | 6-month follow-up
  Use of smoking cessation services will be measured by a self-reported question: Have you ever used smoking cessation services in the past 7 days?
Respiratory symptoms | 3-month follow-up
  Respiratory symptoms will be measured by a self-reported question: Have you ever experienced respiratory symptoms in the past 7 days? If yes, please list.
Respiratory symptoms | 6-month follow-up
  Respiratory symptoms will be measured by a self-reported question: Have you ever experienced respiratory symptoms in the past 7 days? If yes, please list.
Perceived family well-being | 3-month follow-up
  Perceived family well-being will be measured by the Family Apgar Scale. The total scale ranges from 0 to 10, with the higher score indicating a healthier family function.
Perceived family well-being | 6-month follow-up
  Perceived family well-being will be measured by the Family Apgar Scale. The total scale ranges from 0 to 10, with the higher score indicating a healthier family function.
Self-reported life quality | 3-month follow-up
  Quality of life will be measured by the WHOQoL scale. The total score ranges 0 to 100, with higher scores indicates better quality of life.
Self-reported life quality | 6-month follow-up
  Quality of life will be measured by the WHOQoL scale. The total score ranges 0 to 100, with higher scores indicates better quality of life.
Self-reported secondhand exposure | 3-month follow-up
  Self-reported secondhand exposure by children in the past 7 days (yes/no). If yes, we will ask where you are exposed to secondhand smoke and when you are exposed to secondhand smoke.
Self-reported secondhand exposure | 6-month follow-up
  Self-reported secondhand exposure by children in the past 7 days (yes/no). If yes, we will ask where you are exposed to secondhand smoke and when you are exposed to secondhand smoke.
Self-reported thirdhand exposure | 3-month follow-up
  Self-reported thirdhand exposure by children in the past 7 days (yes/no). If yes, we will ask where you are exposed to thirdhand smoke and when you are exposed to thirdhand smoke.
Self-reported thirdhand exposure | 6-month follow-up
  Self-reported thirdhand exposure by children in the past 7 days (yes/no). If yes, we will ask where you are exposed to thirdhand smoke and when you are exposed to thirdhand smoke.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Pokfulam, Hong Kong

IPD SHARING:
Plan to Share IPD: No